CLINICAL TRIAL: NCT00458133
Title: Health Benefits of Aerobic and Resistance Training in Individuals With Type 2 Diabetes
Acronym: HART-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 26046; R01DK068298 (NIH)
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes
Keywords: aerobic exercise; resistance exercise; type 2 diabetes; hemoglobin A1C; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): We randomly assigned 72 individuals to an aerobic exercise training only group.
  Interventions: Behavioral: exercise
- 2 (Experimental): We randomly assigned 73 individuals to an resistance exercise training only group.
  Interventions: Behavioral: exercise
- 3 (Experimental): We randomly assigned 76 individuals to a combination of aerobic plus resistance training group.
  Interventions: Behavioral: exercise
- 4 (Placebo Comparator): We randomly assigned 41 individuals to a stretching and relaxation group.
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — compared effects on HbA1C on aerobic only, resistance only, combination of aerobic and resistance, and a stretching & relaxing groups.

SUMMARY:
The goal of the proposed study, Health Benefits of Aerobic and Resistance Training in individuals with type 2 diabetes (HART-D), is to compare the effect of resistance training alone (RT), resistance in combination with aerobic training (AT+RT), and aerobic training alone (AT) to standard care (SC) on hemoglobin A1C (HbA1C), in initially sedentary women and men with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Although it is generally accepted that regular exercise provides substantial health benefits to individuals with T2D, the exact exercise prescription in terms of type (AT versus RT versus AT+RT) still remains an important research issue, particularly in regard to week-to-week glucose control as assessed by HbA1C.

There is a need for more adequately powered and well-controlled studies to examine the effects of RT, AT and AT+RT on HbA1C in individuals with T2D. With the incidence of T2D expected to increase dramatically in the coming years, it is essential to have a better understanding of the relative benefits of various exercise interventions. This information can help better formulate exercise recommendations for patients with T2D as well as potentially provide more exercise options, which is important given the small percentage of individuals with TD2 who regularly exercise. The study group was sedentary women and men with T2D, aged 30 to 75 years. We randomly assigned 262 individuals to an aerobic exercise training only group (AT; n=72), a resistance training only group (RT; n=73), a combination of aerobic plus resistance training (AT+RT; n=76), or a standard care group (SC; n=41). The AT individuals participated in 3 or 4 training sessions each week for 9 months progressing to a total energy expenditure of 12 kcal/kg/week (KKW), which is an exercise dose consistent with the current public health recommendations for physical activity for individuals with T2D. The target exercise intensity was 50%-80% of baseline VO2 max. The RT group participated in 3 sessions per week (9 exercises, 2-3 sets each), which focuses on large muscle groups. This RT regimen is based on the studies that most successfully improved HbA1C in individuals with T2D. Individuals in the AT+RT group completed 10 KKW of aerobic training and a reduced resistance-training regimen of 2 sessions per week (9 exercises, 1 set of each). The AT+RT regimen represents the exercise recommendations of the American College of Sports Medicine (ACSM) and the American Diabetes Association (ADA).

Simply stated, we compared the effect of resistance training alone, resistance in combination with aerobic training, and aerobic training alone to standard care on HbA1C, in initially sedentary women and men with T2D. The primary outcome measure was HbA1C, an integrated measure of blood glucose control over the past 8-12 weeks. Other outcomes of interest included resting blood pressure, C-reactive protein (CRP), total body fat, and lean muscle mass as measured by DEXA, cardiorespiratory fitness, muscular strength, and metabolic measures including serum cholesterol and triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-75 years
* type 2 diabetes determined by self-report with verification
* 6.5% < HbA1C < 11%
* sedentary lifestyle - not being physically active greater than or equal to 3 days per week for 20 minutes each time for the previous 6 months, and not performing regular resistance exercise

Exclusion Criteria:

* inadequate control of co-morbid conditions
* resting blood pressure greater than or equal to 160/100 mm Hg
* Triglycerides greater than or equal to 500 mg/dL
* BMI is greater than or equal to 48
* current use of an insulin pump or insulin injections other than Lantus
* metal object in the body that may interfere with MRI/MRS scans
* factors that may limit adherence to intervention or affect conduct of the trial

  1. unable or unwilling to communicate with staff, to provide written informed consent, or accept the randomized assignment
  2. failure to complete behavioral run-in and baseline testing
  3. hospitalization for depression in the last 6 months
  4. not physically capable of performing the exercise required for the study protocols
  5. consuming > 14 alcoholic beverages per week
  6. plans to be away > 4 weeks in the next 9 months
  7. lack of support from primary health care provider or family members
  8. significant weight loss in the past year (>20 lbs) or current use of weight loss medications
  9. current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
  10. another member of household is a participant or staff member of HART-D
  11. bariatric surgery
  12. other temporary intervening event, such as sick spouse, bereavement, or recent move
  13. other medical, psychiatric, or behavioral limitations that, in the view of the principal investigator, may interfere with study participation or the ability to follow the intervention protocol
* underlying diseases or conditions likely to limit lifespan and/or affect the safety of the intervention

  1. pregnant or plan on becoming pregnant in the next 9 months
  2. cancers requiring treatment in the past 5 years, unless prognosis is excellent
  3. self-reported HIV or tuberculosis
  4. history or evidence of serious arrythmias, cardiomyopathy, congestive heart failure, aortic aneurysm, or heart transplantation
  5. renal disease: urine dipstick 4+ protein, serum creatinine is greater than or equal to 1.4 mg/dL (women) or is greater than or equal to 1.5 mg/dL (men) or currently receiving dialysis
  6. any other medical condition or disease that is life threatening or that can interfere with or be aggravated by exercise
  7. advanced neuropathy or retinopathy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | at 9 months

SECONDARY OUTCOMES:
Fasting glucose | at 9 months
Basal insulin | at 9 months
Resting blood pressure | at 9 months
C reactive protein | at 9 months
Visceral adiposity | at 9 months
Body Composition | at 9 months
Cardiorespiratory fitness | at 9 months
Muscular strength | at 9 months
metabolic measures, including serum cholesterol and triglycerides | at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Church, MPH, MD, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Zinman B, Ruderman N, Campaigne BN, Devlin JT, Schneider SH; American Diabetes Association. Physical activity/exercise and diabetes mellitus. Diabetes Care. 2003 Jan;26 Suppl 1:S73-7. doi: 10.2337/diacare.26.2007.s73. No abstract available. PMID 12502622
- [Background] Albright A, Franz M, Hornsby G, Kriska A, Marrero D, Ullrich I, Verity LS. American College of Sports Medicine position stand. Exercise and type 2 diabetes. Med Sci Sports Exerc. 2000 Jul;32(7):1345-60. doi: 10.1097/00005768-200007000-00024. PMID 10912903
- [Background] Hamdy O, Goodyear LJ, Horton ES. Diet and exercise in type 2 diabetes mellitus. Endocrinol Metab Clin North Am. 2001 Dec;30(4):883-907. doi: 10.1016/s0889-8529(05)70220-6. PMID 11727404
- [Background] Kelley DE, Goodpaster BH. Effects of exercise on glucose homeostasis in Type 2 diabetes mellitus. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S495-501; discussion S528-9. doi: 10.1097/00005768-200106001-00020. PMID 11427776
- [Background] Nelson KM, Reiber G, Boyko EJ; NHANES III. Diet and exercise among adults with type 2 diabetes: findings from the third national health and nutrition examination survey (NHANES III). Diabetes Care. 2002 Oct;25(10):1722-8. doi: 10.2337/diacare.25.10.1722. PMID 12351468
- [Background] Khaw KT, Wareham N, Luben R, Bingham S, Oakes S, Welch A, Day N. Glycated haemoglobin, diabetes, and mortality in men in Norfolk cohort of european prospective investigation of cancer and nutrition (EPIC-Norfolk). BMJ. 2001 Jan 6;322(7277):15-8. doi: 10.1136/bmj.322.7277.15. PMID 11141143
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Background] Ishii T, Yamakita T, Sato T, Tanaka S, Fujii S. Resistance training improves insulin sensitivity in NIDDM subjects without altering maximal oxygen uptake. Diabetes Care. 1998 Aug;21(8):1353-5. doi: 10.2337/diacare.21.8.1353. PMID 9702447
- [Background] Baldi JC, Snowling N. Resistance training improves glycaemic control in obese type 2 diabetic men. Int J Sports Med. 2003 Aug;24(6):419-23. doi: 10.1055/s-2003-41173. PMID 12905089
- [Background] Castaneda C, Layne JE, Munoz-Orians L, Gordon PL, Walsmith J, Foldvari M, Roubenoff R, Tucker KL, Nelson ME. A randomized controlled trial of resistance exercise training to improve glycemic control in older adults with type 2 diabetes. Diabetes Care. 2002 Dec;25(12):2335-41. doi: 10.2337/diacare.25.12.2335. PMID 12453982
- [Background] Dunstan DW, Daly RM, Owen N, Jolley D, De Courten M, Shaw J, Zimmet P. High-intensity resistance training improves glycemic control in older patients with type 2 diabetes. Diabetes Care. 2002 Oct;25(10):1729-36. doi: 10.2337/diacare.25.10.1729. PMID 12351469
- [Background] Kumar S, Boulton AJ, Beck-Nielsen H, Berthezene F, Muggeo M, Persson B, Spinas GA, Donoghue S, Lettis S, Stewart-Long P. Troglitazone, an insulin action enhancer, improves metabolic control in NIDDM patients. Troglitazone Study Group. Diabetologia. 1996 Jun;39(6):701-9. doi: 10.1007/BF00418542. PMID 8781766
- [Background] Hanley AJ, Williams K, Stern MP, Haffner SM. Homeostasis model assessment of insulin resistance in relation to the incidence of cardiovascular disease: the San Antonio Heart Study. Diabetes Care. 2002 Jul;25(7):1177-84. doi: 10.2337/diacare.25.7.1177. PMID 12087016
- [Background] Katsuki A, Sumida Y, Gabazza EC, Murashima S, Furuta M, Araki-Sasaki R, Hori Y, Yano Y, Adachi Y. Homeostasis model assessment is a reliable indicator of insulin resistance during follow-up of patients with type 2 diabetes. Diabetes Care. 2001 Feb;24(2):362-5. doi: 10.2337/diacare.24.2.362. PMID 11213893
- [Background] Dumortier M, Brandou F, Perez-Martin A, Fedou C, Mercier J, Brun JF. Low intensity endurance exercise targeted for lipid oxidation improves body composition and insulin sensitivity in patients with the metabolic syndrome. Diabetes Metab. 2003 Nov;29(5):509-18. doi: 10.1016/s1262-3636(07)70065-4. PMID 14631328
- [Background] Helge JW. Prolonged adaptation to fat-rich diet and training; effects on body fat stores and insulin resistance in man. Int J Obes Relat Metab Disord. 2002 Aug;26(8):1118-24. doi: 10.1038/sj.ijo.0802058. PMID 12119578
- [Background] Miyatake N, Takahashi K, Wada J, Nishikawa H, Morishita A, Suzuki H, Kunitomi M, Makino H, Kira S, Fujii M. Daily exercise lowers blood pressure and reduces visceral adipose tissue areas in overweight Japanese men. Diabetes Res Clin Pract. 2003 Dec;62(3):149-57. doi: 10.1016/s0168-8227(03)00176-1. PMID 14625129
- [Background] Stewart KJ. Exercise training and the cardiovascular consequences of type 2 diabetes and hypertension: plausible mechanisms for improving cardiovascular health. JAMA. 2002 Oct 2;288(13):1622-31. doi: 10.1001/jama.288.13.1622. PMID 12350193
- [Background] Grossman E, Messerli FH, Goldbourt U. High blood pressure and diabetes mellitus: are all antihypertensive drugs created equal? Arch Intern Med. 2000 Sep 11;160(16):2447-52. doi: 10.1001/archinte.160.16.2447. PMID 10979055
- [Background] Kelley GA, Kelley KA, Tran ZV. Aerobic exercise and resting blood pressure: a meta-analytic review of randomized, controlled trials. Prev Cardiol. 2001 Spring;4(2):73-80. doi: 10.1111/j.1520-037x.2001.00529.x. PMID 11828203
- [Background] Leon AS, Sanchez OA. Response of blood lipids to exercise training alone or combined with dietary intervention. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S502-15; discussion S528-9. doi: 10.1097/00005768-200106001-00021. PMID 11427777
- [Background] Taylor PA, Ward A. Women, high-density lipoprotein cholesterol, and exercise. Arch Intern Med. 1993 May 24;153(10):1178-84. PMID 8494471
- [Background] Durstine JL, Haskell WL. Effects of exercise training on plasma lipids and lipoproteins. Exerc Sport Sci Rev. 1994;22:477-521. No abstract available. PMID 7925552
- [Background] Maiorana A, O'Driscoll G, Goodman C, Taylor R, Green D. Combined aerobic and resistance exercise improves glycemic control and fitness in type 2 diabetes. Diabetes Res Clin Pract. 2002 May;56(2):115-23. doi: 10.1016/s0168-8227(01)00368-0. PMID 11891019
- [Background] Dunstan DW, Puddey IB, Beilin LJ, Burke V, Morton AR, Stanton KG. Effects of a short-term circuit weight training program on glycaemic control in NIDDM. Diabetes Res Clin Pract. 1998 Apr;40(1):53-61. doi: 10.1016/s0168-8227(98)00027-8. PMID 9699091
- [Background] Eriksson J, Taimela S, Eriksson K, Parviainen S, Peltonen J, Kujala U. Resistance training in the treatment of non-insulin-dependent diabetes mellitus. Int J Sports Med. 1997 May;18(4):242-6. doi: 10.1055/s-2007-972627. PMID 9231838
- [Background] Honkola A, Forsen T, Eriksson J. Resistance training improves the metabolic profile in individuals with type 2 diabetes. Acta Diabetol. 1997 Dec;34(4):245-8. doi: 10.1007/s005920050082. PMID 9451466
- [Background] Haffner SM. Insulin resistance, inflammation, and the prediabetic state. Am J Cardiol. 2003 Aug 18;92(4A):18J-26J. doi: 10.1016/s0002-9149(03)00612-x. PMID 12957323
- [Background] Ridker PM, Hennekens CH, Buring JE, Rifai N. C-reactive protein and other markers of inflammation in the prediction of cardiovascular disease in women. N Engl J Med. 2000 Mar 23;342(12):836-43. doi: 10.1056/NEJM200003233421202. PMID 10733371
- [Background] Ridker PM. High-sensitivity C-reactive protein: potential adjunct for global risk assessment in the primary prevention of cardiovascular disease. Circulation. 2001 Apr 3;103(13):1813-8. doi: 10.1161/01.cir.103.13.1813. PMID 11282915
- [Background] Church TS, Barlow CE, Earnest CP, Kampert JB, Priest EL, Blair SN. Associations between cardiorespiratory fitness and C-reactive protein in men. Arterioscler Thromb Vasc Biol. 2002 Nov 1;22(11):1869-76. doi: 10.1161/01.atv.0000036611.77940.f8. PMID 12426218
- [Background] Nguyen-Duy TB, Nichaman MZ, Church TS, Blair SN, Ross R. Visceral fat and liver fat are independent predictors of metabolic risk factors in men. Am J Physiol Endocrinol Metab. 2003 Jun;284(6):E1065-71. doi: 10.1152/ajpendo.00442.2002. Epub 2003 Jan 28. PMID 12554597
- [Background] Mourier A, Gautier JF, De Kerviler E, Bigard AX, Villette JM, Garnier JP, Duvallet A, Guezennec CY, Cathelineau G. Mobilization of visceral adipose tissue related to the improvement in insulin sensitivity in response to physical training in NIDDM. Effects of branched-chain amino acid supplements. Diabetes Care. 1997 Mar;20(3):385-91. doi: 10.2337/diacare.20.3.385. PMID 9051392
- [Background] Kohl HW 3rd, Dunn AL, Marcus BH, Blair SN. A randomized trial of physical activity interventions: design and baseline data from project active. Med Sci Sports Exerc. 1998 Feb;30(2):275-83. doi: 10.1097/00005768-199802000-00016. PMID 9502357
- [Background] Blair SN, Applegate WB, Dunn AL, Ettinger WH, Haskell WL, King AC, Morgan TM, Shih JA, Simons-Morton DG. Activity Counseling Trial (ACT): rationale, design, and methods. Activity Counseling Trial Research Group. Med Sci Sports Exerc. 1998 Jul;30(7):1097-106. doi: 10.1097/00005768-199807000-00012. PMID 9662679
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Smutok MA, Reece C, Kokkinos PF, Farmer C, Dawson P, Shulman R, DeVane-Bell J, Patterson J, Charabogos C, Goldberg AP, et al. Aerobic versus strength training for risk factor intervention in middle-aged men at high risk for coronary heart disease. Metabolism. 1993 Feb;42(2):177-84. doi: 10.1016/0026-0495(93)90032-j. PMID 8474314
- [Background] Smutok MA, Reece C, Kokkinos PF, Farmer CM, Dawson PK, DeVane J, Patterson J, Goldberg AP, Hurley BF. Effects of exercise training modality on glucose tolerance in men with abnormal glucose regulation. Int J Sports Med. 1994 Aug;15(6):283-9. doi: 10.1055/s-2007-1021061. PMID 7822064
- [Background] Physical activity and cardiovascular health. NIH Consensus Development Panel on Physical Activity and Cardiovascular Health. JAMA. 1996 Jul 17;276(3):241-6. PMID 8667571
- [Background] Surgeon General's report on physical activity and health. From the Centers for Disease Control and Prevention. JAMA. 1996 Aug 21;276(7):522. No abstract available. PMID 8709391
- [Background] Snyder KA, Donnelly JE, Jabobsen DJ, Hertner G, Jakicic JM. The effects of long-term, moderate intensity, intermittent exercise on aerobic capacity, body composition, blood lipids, insulin and glucose in overweight females. Int J Obes Relat Metab Disord. 1997 Dec;21(12):1180-9. doi: 10.1038/sj.ijo.0800533. PMID 9426387
- [Background] Willey KA, Singh MA. Battling insulin resistance in elderly obese people with type 2 diabetes: bring on the heavy weights. Diabetes Care. 2003 May;26(5):1580-8. doi: 10.2337/diacare.26.5.1580. PMID 12716822
- [Result] Church TS, Blair SN, Cocreham S, Johannsen N, Johnson W, Kramer K, Mikus CR, Myers V, Nauta M, Rodarte RQ, Sparks L, Thompson A, Earnest CP. Effects of aerobic and resistance training on hemoglobin A1c levels in patients with type 2 diabetes: a randomized controlled trial. JAMA. 2010 Nov 24;304(20):2253-62. doi: 10.1001/jama.2010.1710. PMID 21098771
- [Result] Swift DL, Johannsen NM, Earnest CP, Blair SN, Church TS. Effect of exercise training modality on C-reactive protein in type 2 diabetes. Med Sci Sports Exerc. 2012 Jun;44(6):1028-34. doi: 10.1249/MSS.0b013e31824526cc. PMID 22157880
- [Result] Swift DL, Johannsen NM, Myers VH, Earnest CP, Smits JA, Blair SN, Church TS. The effect of exercise training modality on serum brain derived neurotrophic factor levels in individuals with type 2 diabetes. PLoS One. 2012;7(8):e42785. doi: 10.1371/journal.pone.0042785. Epub 2012 Aug 6. PMID 22880108
- [Derived] Senechal M, Johannsen NM, Swift DL, Earnest CP, Lavie CJ, Blair SN, Church TS. Association between Changes in Muscle Quality with Exercise Training and Changes in Cardiorespiratory Fitness Measures in Individuals with Type 2 Diabetes Mellitus: Results from the HART-D Study. PLoS One. 2015 Aug 7;10(8):e0135057. doi: 10.1371/journal.pone.0135057. eCollection 2015. PMID 26252477
- [Derived] Pandey A, Swift DL, McGuire DK, Ayers CR, Neeland IJ, Blair SN, Johannsen N, Earnest CP, Berry JD, Church TS. Metabolic Effects of Exercise Training Among Fitness-Nonresponsive Patients With Type 2 Diabetes: The HART-D Study. Diabetes Care. 2015 Aug;38(8):1494-501. doi: 10.2337/dc14-2378. Epub 2015 Jun 17. PMID 26084342
- [Derived] Henagan TM, Stewart LK, Forney LA, Sparks LM, Johannsen N, Church TS. PGC1alpha -1 Nucleosome Position and Splice Variant Expression and Cardiovascular Disease Risk in Overweight and Obese Individuals. PPAR Res. 2014;2014:895734. doi: 10.1155/2014/895734. Epub 2014 Dec 28. PMID 25614734
- [Derived] Johannsen NM, Swift DL, Lavie CJ, Earnest CP, Blair SN, Church TS. Categorical analysis of the impact of aerobic and resistance exercise training, alone and in combination, on cardiorespiratory fitness levels in patients with type 2 diabetes: results from the HART-D study. Diabetes Care. 2013 Oct;36(10):3305-12. doi: 10.2337/dc12-2194. Epub 2013 Jul 22. PMID 23877979
- [Derived] Johannsen NM, Sparks LM, Zhang Z, Earnest CP, Smith SR, Church TS, Ravussin E. Determinants of the Changes in Glycemic Control with Exercise Training in Type 2 Diabetes: A Randomized Trial. PLoS One. 2013 Jun 21;8(6):e62973. doi: 10.1371/journal.pone.0062973. Print 2013. PMID 23805175
- [Derived] Senechal M, Swift DL, Johannsen NM, Blair SN, Earnest CP, Lavie CJ, Church TS. Changes in body fat distribution and fitness are associated with changes in hemoglobin A1c after 9 months of exercise training: results from the HART-D study. Diabetes Care. 2013 Sep;36(9):2843-9. doi: 10.2337/dc12-2428. Epub 2013 May 13. PMID 23670995